CLINICAL TRIAL: NCT07387692
Title: Randomized Controlled Trial of Peer Support for Whole Health
Brief Title: Peer Support for Whole Health for Veterans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RRD4-011-25M; 1I01RD000397-01A (Other Grant/Funding Number: VA ORD)
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Psychosocial Functioning; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer Support for Whole Health (Experimental): In this arm, Veteran participants will receive Peer Support for Whole Health from VA peer support staff.
  Interventions: Behavioral: Peer Support for Whole Health
- Self-Directed Whole Health (Active Comparator): In this arm, Veteran participants will receive information about Whole Health tools and resources from research staff.
  Interventions: Behavioral: Self-Directed Whole Health

INTERVENTIONS:
Behavioral: Peer Support for Whole Health — Veteran participants have one-on-one appointments with VA peer support staff to talk about VA Whole Health including goals and progress.
  Arms: Peer Support for Whole Health
Behavioral: Self-Directed Whole Health — Veteran participants have an appointment with research staff and receive information about VA Whole Health tools and resources including handouts, websites, and apps.
  Arms: Self-Directed Whole Health

SUMMARY:
This project is evaluating a new intervention, Peer Support for Whole Health. Peer Support for Whole Health is delivered by peer support specialists, Veterans who are in recovery from mental health or substance use concerns who are employed to help other Veterans. Peer Support for Whole Health uses the Whole Health model to talk about values and self-care in all areas of life. Peer Support for Whole Health is designed to help Veterans who have difficulty with their relationships, work, or day-to-day life and may have behavioral health concerns. Peer Support for Whole Health is designed for Veterans in primary care who are not engaged in mental health or substance use treatment. The goal of this study is to find out whether Peer Support for Whole Health helps Veterans with relationships, work, or day-to-day life. This project will also study whether Peer Support for Whole Health improves well-being and mental health. Finally, this study will seek to understand how Peer Support for Whole Health works and which Veterans it helps the most.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* enrolled in primary care at one of the study sites
* have some challenges with day-to-day life (e.g., relationships, work, school, getting things done) based on a standard questionnaire
* have a recent primary care medical record note documenting potential behavioral health concerns or symptoms
* fully understand the research study

Exclusion Criteria:

* not be enrolled in current peer support services, mental health services, or other similar services
* at risk for suicide or other high-risk concerns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2027-01-04 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Inventory of Psychosocial Functioning | 9 months
  The Inventory of Psychosocial Functioning measures all key areas of psychosocial functioning including social functioning (e.g., family, parenting, romantic relationships, friendships), vocational functioning (e.g., work and school), and self-care (e.g., chores, diet, medical care).

SECONDARY OUTCOMES:
Well-Being Signs | 9 months
  The Well-Being Signs assess satisfaction, involvement, and functioning in important aspects of life.
Depression Anxiety and Stress Scales (DASS-21) | 9 months
  The Depression Anxiety and Stress Scales-21 assess psychological distress including anxiety, depression, and stress-related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Emily M. Johnson, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (2):
- United States (2):
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymous, de-identified data can be made available upon reasonable written request following conclusion of the trial. All identifiable information will be removed prior to sharing, and the minimum amount of data required to achieve the purposes of the request will be shared.